CLINICAL TRIAL: NCT00832546
Title: A Double-Blind, Randomized, Placebo Controlled, Cross-Over, Safety Tolerance and Experimental Hyperalgesia Study of Oral NGX426 in Healthy Male Volunteers
Brief Title: A Safety Tolerance and Experimental Hyperalgesia Study of Oral NGX426 in Healthy Male Voluneteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TorreyPines Therapeutics (Industry)
Responsible Party: Susan Mellberg, R.N., M.B.A.; VP, Project Management, TorreyPines Therapeutics, Inc.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NGX426CLP1003
Record Dates: First submitted 2009-01-28; First posted 2009-01-30 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Healthy; Hyperalgesia
MeSH Terms: conditions — Hyperalgesia | interventions — Powders; Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Experimental): Powder in solution
  Interventions: Drug: Oral NGX426 (Powder in solution)
- 3 (Experimental)
  Interventions: Drug: Oral NGX426 (Powder in solution)

INTERVENTIONS:
Drug: Placebo
  Arms: 1
Drug: Oral NGX426 (Powder in solution)
  Arms: 2; 3

SUMMARY:
The purpose of this study is to determine the effects of NGX426 on intradermal capsaicin induced pain in hyperalgesia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males, age 21-55

Exclusion Criteria:

* Allergy to study drug

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wallace, M.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, California, United States